CLINICAL TRIAL: NCT01694836
Title: Multicenter, Placebo-controlled, Long-term Study of Depigoid Birch 5000 in Adults and Adolescents With Allergic Rhinitis and/or Rhinoconjunctivitis With or Without Intermittent Asthma
Brief Title: Depigoid Birch 5000 Longterm Study in Adults and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leti Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 603-PG-PSC-191; 2012-000414-11 (EudraCT Number)
Record Dates: First submitted 2012-08-27; First posted 2012-09-27 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinitis/Rhinoconjunctivitis +-Intermittent Asthma; Sensitization Against Betula Alba (Birch) Pollen
Keywords: Allergic rhinitis; Allergic rhinoconjunctivitis; Allergy induced asthma; Birch (Betula alba); Hayfever; Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depigoid Birch 5.000 DPP/ml (Experimental): Suspension for s.c. injection. Treatment schedule:
  1. Build-up phase (1 day: 0,2 ml+0,3 ml at interval of 30 minutes)
  2. Maintenance phase (3 years: 0,5 ml at intervals of 4-6 weeks)
  Interventions: Biological: s.c. injection
- Placebo (Placebo Comparator): Suspension for s.c. injection. Treatment schedule:
  1. Build-up phase (1 day: 0,2 ml+0,3 ml at interval of 30 minutes)
  2. Maintenance phase (3 years: 0,5 ml at intervals of 4-6 weeks)
  Interventions: Biological: s.c. injection

INTERVENTIONS:
Biological: s.c. injection — 3 years of therapy followed by 2 years (seasons) of treatment-free observational period
  Other Names: Depigoid(R)Birch

SUMMARY:
Specific immunotherapy for IgE mediated sensitization to birch pollen. Long-term study to assess safety and efficacy of Depigoid(R)Birch 5000 - a modified pollen extract of Betula alba (Birch) - versus placebo.

DETAILED DESCRIPTION:
Investigation of the long-term efficacy and safety of Depigoid Birch 5000 according to the perennial treatment regimen in comparison to placebo in adult and adolescent patients with birch pollen-induced allergic rhinitis and/or rhinoconjunctivitis to show superiority vs. placebo.

As the study includes adolescent patients it is run under an approved PIP.

Total study duration per patient will be 5 years: 3 years of perennial treatment (application of study medication at intervals of 4-6 weeks) followed by a treatment-free observational phase of 2 years (seasons).

ELIGIBILITY:
Inclusion Criteria:

* Availability of an appropriately signed and dated informed consent before any study specific examination,
* Clinical history of at least 2 years of seasonal allergic rhinitis and/or rhinoconjunctivitis with or without intermittent asthma due to birch pollen allergy that has required repeated use of symptomatic treatment,
* Patients must have a minimum level of perception of symptoms from previous seasons defined as at least a moderate symptom level (i.e. a score of 2 on the 4-point-Likert scale) in at least 2 symptom categories prior to randomization,
* Lung function ≥ 80% of the predicted normal value,
* IgE-mediated sensitization has to be verified by:

  * suggestive medical history, and
  * specific IgE reactivity to birch pollen (CAP-RAST ≥ 2), and
  * a positive SPT to birch pollen at screening or within 1 months prior to the screening visit. An SPT is considered positive if it results in a wheal diameter of at least 3.0 mm
* Internet access so that patients can complete the eDiary daily via internet during all 5 pollen seasons covered by the study protocol.

Exclusion Criteria:

* History of significant clinical manifestations of allergy as a result of sensitization against co-allergies, particularly-but not limited to-grass or weed pollen and perennial allergens (e.g. house dust mites, cat or dog).
* History of anaphylactic reaction.
* Moderate or severe persistent asthma (GINA 3 or 4).
* Mild persistent asthma (GINA 2), according to the Global Initiative for Asthma Guidelines, necessitating treatment with inhaled glucocorticoids at a daily dose level of > 400 µg budesonide dose equivalents.
* Lung function < 80% of the predicted normal value (for PEF: highest result of 3 measurements).
* Acute or chronic inflammatory or infectious airway diseases including recurrent acute or chronic sinusitis.
* Chronic structural diseases of the affected organs (e.g. eye, nose, lung).
* History or presence of confirmed or potential diseases of the immune system including autoimmune diseases and immune deficiencies of actual clinical relevance.
* Any disease that prohibits the use of adrenaline (e.g. hyperthyroidism).
* Atopic dermatitis with SCORAD >30 in the past or at screening.
* Ongoing or past full courses of SIT against birch pollen within the last 5 years.
* Topical and systemic treatment with β-blockers.
* Concomitant treatment with substances interfering with the immune system beginning 1 week prior to start of treatment.
* Use of systemic corticosteroids within 3 months prior to Visit 1-1.
* Immunization with vaccines within 7 days prior to Visit 1-1.
* Treatment with antihistamines for any reason other than allergic symptoms due to birch pollen allergy.
* Changed residence between geographical regions since the last birch pollen season or not staying in the geographical region during the pre-determined birch pollen season.
* Nursing (lactating) women or women with a positive pregnancy test at the screening visit. Women of childbearing potential must be using highly effective contraception during participation in this clinical study. A highly effective method of birth control is defined as one that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, or vasectomised partner.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Proof of efficacy (superiority vs. placebo) by means of the combined Symptom and Medication Score (SMS). | after 5 years
  For the primary outcome the SMS of nasal and ocular symptoms and their respective Rescue Medication score is used to assess efficacy of the perennial treatment regimen of Depigoid Birch 5000 DPP/mL versus placebo after 5 years (comprising 3 years of treatment plus 2 years treatment-free follow-up). An interim analysis will be conducted after 2 years.
  Data are captured via eDiary to be completed by the patients during each of the 5 pollen seasons within the duration of the study, starting prior to onset of pollen flight until after the end of the pollen seasons.

SECONDARY OUTCOMES:
Symptom score (SS) during the 1st, 3rd, and 4th pollen seasons. | after 1 year, 2 years, 3 years, 4 years and 5 years
  Differences between treatment groups also including pulmonary symptoms and for asthmatic/non-asthmatic patients.
  Data are captured via eDiary to be completed by the patients during each of the 5 pollen seasons within the duration of the study, starting prior to onset of pollen flight until after the end of the pollen seasons.
Rescue Medication Score (RMS) during the 1st, 3rd, and 4th pollen season (futility and interim analyses). | after 1 year, 2 years, 3 years, 4 years and 5 years
  Differences between treatment groups also including pulmonary symptoms and for asthmatic/non-asthmatic patients.
  Data are captured via eDiary to be completed by the patients during each of the 5 pollen seasons within the duration of the study, starting prior to onset of pollen flight until afte the end of the pollen seasons.
combined Symptoms and Rescue Medication Score (SMS) during the 1st, 3rd, and 4th pollen season including pulmonary symptoms. | after 1 year, 2 years, 3 years and 4 years
  Differences between treatment groups, during all 5 pollen seasons also including pulmonary symptoms and for asthmatic/non-asthmatic patients.
  Data are captured via eDiary to be completed by the patients during each of the 5 pollen seasons within the duration of the study, starting prior to onset of pollen flight until after the end of the pollen seasons.
Rhinitis Quality of Life Questionnaire (RQLQ) resp. RQLQ for adolescent patients (AdolRQLQ) | Screening and after 1 year, 2 years, 3 years, 4 years and 5 years
  Changes to baseline and difference between treatment groups during all 5 pollen seasons
Immunology parameters (Total IgE, specific IgE, specific IgG1 and IgG4) | Screening, after years 1, 2, 3 and 5 (resp. end of study)
  Differences within patients and between treatment groups
Disease modifying effect after 5 years | after 5 years
  Difference between treatment groups. Incidence of asthma and new sensitizations.
Clinical chemistry: Number of patients with outside range values | Screening, after years 2, 3 and 5
  Differences between treatment groups
Adverse events: number of patients with AEs/SAEs | throughout the whole study duration
  Including symptoms reported by patients in eDiary. Differences between treatment groups including but not limited to differences in severity levels of systemic reactions (SRs), immediate and local reaction including calculation of ratios per injection
Serum levels of Aluminium hydroxide (Pharmacokinetics) | prior and after 1st and 2nd application of IMP and after 1 year
  Serum Aluminium hydroxide levels are assessed in a subgroup of 24 patients. Differences between treatment groups (adult patients only) Sampling: prior to 1st application of IMP, 4 time points after 1st, 2nd and 10th application (after 1 year). 24 hrs. urine at these 3 time points
Vitamin D3 level | baseline and end of study
  Possible influence on specific immunotherapy. Exploratory evaluation
Hematology: Number of patients with outside range values | Screening, after years 2, 3 and 5
  Differences between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Natalja Novak, Prof. Dr., Principal Investigator — Klinik für Dermatologie und Allergologie der Universität Bonn; Angelika Sager, Dr. med., Study Director — Leti Pharma GmbH
Locations (2):
- Germany (2):
  - Hautarztpraxis, Berlin
  - Klinik und Poliklinik für Dermatologie und Allergologie der Universität, Bonn